CLINICAL TRIAL: NCT03142815
Title: Correlation Between Arterial Stiffness and Aortic-to-radial Pressure Gradient After Cardiopulmonary Bypass
Brief Title: Aortic-Radial Pressure Gradients Post CPB
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Kenichi Ueda, Clinical Associate Professor, University of Iowa
Other Study IDs: 201703834
Record Dates: First submitted 2017-04-28; First posted 2017-05-05 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Bypass Graft (CABG), Arterial stiffness
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will examine whether pre-operative, non-invasive arterial stiffness measurements can be used to predict which patients will develop an aortic-to-radial pressure gradient after coronary artery bypass graft (CABG) surgery. A previous small study by Kanazawa, et al. demonstrated in patients who developed an aortic-to-radial pressure gradient after CABG surgery, the pulse wave velocity (PWV) was higher in the aorta and decreased when moving toward the radial artery. In the patients who did not develop a pressure gradient, the PWV started lower in the aorta and increased when moving towards the periphery.

The purpose of this investigation is to examine whether pre-operative PWV measurements can be used to identify patients who will develop an aortic to radial pressure gradient after CABG surgery.

Applanation tonometry will be performed on the right carotid and femoral arteries to assess carotid-femoral pulse wave velocity, a surrogate for aortic stiffness. (SphygmoCor system, AtCor Medical, Sydney, Australia). The measurement will be obtained before induction of general anesthesia in the presurgical area. Also in the presurgical area, a non-invasive cardiac output (CO) measurement will be obtained by using the ICON Device (Osypka Medical, La Jolla, California). This CO value will be used to compare to the CO values obtained invasively in the operating room.

DETAILED DESCRIPTION:
The purpose of the study is determine if there is a relationship between pre-operative vascular characteristics including, carotid-femoral pulse wave velocity (cfPWV), Augmentation Index(AI) and central aortic pressure, and the development of a pressure gradient between the aorta and radial artery after cardiopulmonary bypass.

The procedures necessary to achieve the desired outcomes are as follows. The first measurement made by the research team will be pre-operative cardiac output (CO) measurement. The ICON device is a non-invasive device that measures CO, or the amount of blood that your heart pumps per minute. This device utilizes four stickers that are attached to skin, two on the left side of the neck and two located on the left side of the chest. These stickers function similarly to electrocardiogram (EKG) stickers that measure the electrical activity of your heart. After attachment of the stickers, the ICON device will be used to make a measurement of CO, which takes 1-2 minutes. After the measurement, the stickers will be removed and the ICON device will not be used again in the study.

Secondly, pre-operative cfPWV, AI, and central aortic pressure measurements will be made. The Sphygmocor device will be utilized to make the pre-operative cfPWV, AI and central aortic pressure measurements. First, the AI measurements will be made using a non-invasive blood pressure cuff placed on the right arm. The patient's blood pressure will be measured twice in a row with this special blood pressure cuff. The blood pressure cuff on the right arm will be removed and then a cuff will be placed around the right thigh. Measurements will be made with a paper ruler from the patient's neck to the cuff on their leg. To make the cfPWV measurements, the cuff on the thigh will inflate while a pressure probe will be placed on the skin of the patient's right neck. Four measurements of cfPWV will be made with this technique.

The intraoperative central aortic pressure measurement will be accomplished with the help of the cardiothoracic surgeon. The surgeon will place a catheter in the aorta as part of the coronary artery bypass grafting surgery. This catheter will be connected to the artificial heart-lung machine. Prior to turning on the heart-lung machine, the pressure in the aorta will be measured with this catheter. This is the standard of care for this type of surgery and will not delay the surgery. After the artificial heart-lung machine is turned off but before the catheter is removed from the aorta, the pressure will once again be measured.

In order to measure intraoperative CO values, we will utilize the pulmonary artery (PA) catheter that was placed at the beginning of the surgery.. The patient will have a catheter placed in the right side of the neck that will travel through the heart and into a branch of the artery that goes from the heart to the lungs. This catheter will have the ability to measure the amount of blood that is pumped from the heart per minute. At the same times that the pressure in the aorta is measured (as above), the amount of blood that is pumped from the heart per minute will be measured.

Lastly measurement of peripheral artery blood pressure will be accomplished with a right radial arterial catheter. Prior to the start of surgery, the patient will receive a special catheter in the radial artery of their right arm. This is the standard of care for blood pressure monitoring in this type of surgery. At the same times during the surgery that the pressure is being measured from the aortic catheter, the pressure will be measured from the catheter in the right radial artery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age 40-80, who are scheduled to undergo elective coronary artery bypass graft (CABG) surgery at the University of Iowa Hospitals and Clinics.

Exclusion Criteria:

* off-pump CABG surgery, emergency cases, patients who already have a balloon pump or major valvular heart disease, and if preoperative PWV is not obtainable for any reason.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients aged 40-80 years old who are scheduled to undergo elective on-pump coronary artery bypass graft (CABG) surgery.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Comparison of pre-operative carotid-femoral pulse wave velocity (cfPWV)between patients who develop an aortic-to-radial pressure gradient after coronary artery bypass surgery and those who don't develop a pressure gradient | 1 day (day of surgery)
  The study is aimed to compare cfPWV between patients who develop an aortic-to-radial pressure gradient after coronary artery bypass and those who don't who are undergoing coronary artery bypass graft surgery. Arterial stiffness will be measured by pulse wave velocity (m/s) with a SphygmoCor® device (Atcor, Sydney, Australia)
Comparison of AI between patients who develop an aortic-to-radial pressure gradient and those who don't a pressure gradient | 1 day (day of surgery)
  The study is aimed to compare AI between patients who develop an aortic-to-radial pressure gradient after coronary artery bypass and those who don't who are undergoing coronary artery bypass graft surgery. Arterial stiffness will be measured by pulse wave velocity (m/s) with a SphygmoCor® device

SECONDARY OUTCOMES:
Aortic pressure | 1 day (day of surgery)
  Central aortic pressure will be measured before and after bypass.
Pulse pressure | 1 day (day of surgery)
  Pulse pressure will be measured.
CO | 1 day (day of surgery)
  Cardiac Output before and after coronary artery bypass
SVR | 1 day (day of surgery)
  Systemic vascular resistance before and after coronary artery bypass
Risk factors | 1 day (day of surgery)
  Pre-operative risk factors will be examined for any indication of development of aortic-to-radial pressure gradient after coronary artery bypass graft surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Ueda, MD, PhD, Principal Investigator — University of Iowa Department of Anesthesia
Locations (1):
- University of Iowa Hosptials and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan currently to share IPD with other researchers.

REFERENCES:
- [Background] Kanazawa M, Fukuyama H, Kinefuchi Y, Takiguchi M, Suzuki T. Relationship between aortic-to-radial arterial pressure gradient after cardiopulmonary bypass and changes in arterial elasticity. Anesthesiology. 2003 Jul;99(1):48-53. doi: 10.1097/00000542-200307000-00011. PMID 12826841
- [Background] O'Rourke MF, Nichols WW. Aortic diameter, aortic stiffness, and wave reflection increase with age and isolated systolic hypertension. Hypertension. 2005 Apr;45(4):652-8. doi: 10.1161/01.HYP.0000153793.84859.b8. Epub 2005 Feb 7. No abstract available. PMID 15699456
- [Background] Schmidt C, Theilmeier G, Van Aken H, Korsmeier P, Wirtz SP, Berendes E, Hoffmeier A, Meissner A. Comparison of electrical velocimetry and transoesophageal Doppler echocardiography for measuring stroke volume and cardiac output. Br J Anaesth. 2005 Nov;95(5):603-10. doi: 10.1093/bja/aei224. Epub 2005 Sep 9. PMID 16155037
- [Background] Zoremba N, Bickenbach J, Krauss B, Rossaint R, Kuhlen R, Schalte G. Comparison of electrical velocimetry and thermodilution techniques for the measurement of cardiac output. Acta Anaesthesiol Scand. 2007 Nov;51(10):1314-9. doi: 10.1111/j.1399-6576.2007.01445.x. PMID 17944633